CLINICAL TRIAL: NCT02756208
Title: A Phase I Safety and Immunogenicity Trial of IHV01 in HIV-1 Uninfected Volunteers
Brief Title: A Safety and Immunogenicity Trial of IHV01
Acronym: FLSC-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Auro Vaccines LLC (Industry)
Responsible Party: Principal Investigator, Mohammad Sajadi, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HP-00065547
Record Dates: First submitted 2016-04-17; First posted 2016-04-29 (Estimated); Results first posted 2021-11-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: HIV Infection
Keywords: vaccine; healthy volunteer
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (4):
- 300 ug FLSC vaccine (Experimental): Subjects will be vaccinated with 300 ug FLSC vaccine (highest vaccine dose) on study days 0, 28, 56 and 168.
  Interventions: Biological: 300 ug FLSC vaccine
- 150 ug FLSC vaccine (Experimental): Subjects will be vaccinated with 150 ug FLSC vaccine (middle vaccine dose) on study days 0, 28, 56 and 168.
  Interventions: Biological: 150 ug FLSC vaccine
- 75 ug FLSC vaccine (Experimental): Subjects will be vaccinated with 75 ug FLSC vaccine (lowest vaccine dose) on study days 0, 28, 56 and 168.
  Interventions: Biological: 75 ug FLSC vaccine
- Placebo (Placebo Comparator): Subjects will be vaccinated with placebo (control group) on study days 0, 28, 56 and 168.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: 300 ug FLSC vaccine — FLSC vaccine 300 ug (1.0 mL) given by intramuscular injection into the arm on study Days 0, 28, 56, 168
  Other Names: Full length single chain gp120-CD4 complex vaccine
  Arms: 300 ug FLSC vaccine
Biological: 150 ug FLSC vaccine — FLSC vaccine 150 ug (0.5 mL) given by intramuscular injection into the arm on study Days 0, 28, 56, 168
  Other Names: Full length single chain gp120-CD4 complex vaccine
  Arms: 150 ug FLSC vaccine
Biological: 75 ug FLSC vaccine — FLSC vaccine 75 ug (0.25 mL) given by intramuscular injection into the arm on study Days 0, 28, 56, 168
  Other Names: Full length single chain gp120-CD4 complex vaccine
  Arms: 75 ug FLSC vaccine
Biological: Placebo — Placebo sterile saline (0.25 - 1.0 mL) given by intramuscular injection into the arm on study Days 0, 28, 56, 168
  Other Names: sterile saline
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety of the FLSC vaccine and will be a randomized, placebo-controlled, modified double-blinded dose escalation study in 60 healthy adult volunteers (Human Immunodeficiency Virus-1 uninfected).

DETAILED DESCRIPTION:
This is a Phase 1 randomized, placebo-controlled, modified double-blinded dose escalation study in 60 healthy adult volunteers who are Human Immunodeficiency Virus-1 (HIV-1) uninfected. Participants in the study will receive 4 injections at 0, 4, 8 and 24 weeks and will be followed for an additional 24 weeks. The total study duration will be 48 weeks. As this is a Phase 1 trial, the primary objective is to document safety of the Full Length Single Chain (FLSC) gp120-CD4 complex vaccine with a secondary objective to evaluate immune responses induced by the vaccine. This vaccine is being evaluated as it is constructed so that the gp120 and CD4 moieties form a stable intra-chain binding interaction that forms a transition state structure that presents conserved, conformational domains involved in the early HIV replication process. It is hypothesized that antibodies directed to these epitopes would be highly cross-reactive and potentially useful for HIV vaccine development.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 45 years of age.
2. Sex: Male or Female (female volunteers of child bearing potential must have a negative serum beta human chorionic gonadotropin (b-HCG or pregnancy) test at time of screening and entry into the study and provide assurance of the use of effective(as judged by the investigator) birth control methods or abstinence beginning at least 60 days prior to the study and during the study
3. Documented HIV-1 negative by ELISA
4. Be in good general health without clinically significant medical history, physical examination findings, or clinically significant abnormal laboratory results (i.e., chronic medical conditions as noted in the exclusion criteria such as cancer as well as any conditions that in the opinion of the investigator might pose a risk to the volunteer)
5. No identifiable risk factor for acquisition of HIV infection (i.e., intravenous drug use/needle sharing, unprotected sex with multiple partners)
6. Negative b-HCG pregnancy test on the day of initial vaccination.
7. Negative screen for Hepatitis B surface antigen (HBsAg);
8. Negative screen for antibodies to Hepatitis C virus (Patient may enroll if patient can provide documentation of negative hepatitis C viral load.)
9. Participant must have a CD4 count ( a type of white blood cells) within the normal range of the clinical laboratory utilized for the study and a CD4 percentage within 20% of the normal range of the clinical laboratory
10. Laboratory parameters must be within pre-specified limits as defined by exclusion criteria.
11. Volunteers must be willing and able to provide written informed consent to participate in the study.
12. Available for at least 48 weeks of follow-up.

Exclusion Criteria:

1. High risk behavior for acquisition of HIV within 24 weeks of study entry(i.e., intravenous drug use/needle sharing, unprotected sex with multiple partners)
2. Volunteers with an acute and clinically significant medical event (as determined by the investigator) within the past 30 days of screening.
3. Have active tuberculosis or other systemic infectious process by review of systems and physical examination
4. Have a history of immunodeficiency, autoimmune disease, or use of immunosuppressive medications
5. Current treatment for malignancy other than basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
6. Is pregnant
7. History of any chronic illness that would interfere with conduct or completion of study(as determined by the investigator)
8. Have evidence of psychiatric, medical and/or substance abuse problems during the past 24 weeks that the investigator believes would adversely affect the volunteer's ability to participate in the trial
9. Have occupational or other responsibilities that would prevent completion of participation in the study
10. Have received any live, attenuated vaccine except rabies vaccine within 60 days of study entry
11. Vaccine (FDA approved; e.g. influenza, pneumovax, etc) administration within 30 days of immunization with the study vaccine. NOTE: Medically indicated subunit or killed vaccines (e.g., Hepatitis A or Hepatitis B) should be given prior to trial initiation or after completion of the study immunizations. If patient requires immunization, injections should be given more than 2 weeks prior or 2 weeks after study immunization
12. Have used experimental therapeutic agents within 30 days of study entry
13. Have received blood products or immunoglobulins in the past 12 weeks
14. Have a history of anaphylaxis or other serious adverse reactions to vaccines
15. Have previously received an HIV vaccine
16. Volunteers with any of the following laboratory parameters at the screening visit (within 30 days of immunization): Hemoglobin <10 (without having received a blood or red blood cell transfusion within 30 days prior to laboratory test); neutrophil count <750 cells/mm3; platelet count <50,000/mm3; serum creatinine > 2.0 mg/dL; aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the upper limits of normal; total bilirubin > 1.5 mg/dL
17. Pregnant women or women who are breast-feeding; female volunteers of childbearing potential who are not using or willing to use an effective (as judged by the investigator) barrier contraceptive methods or abstinence while enrolled in this study.
18. Use of any immune modulators or suppressors within 45 days of study entry including but not limited to agents such as interleukins (e.g. IL-2), interferons (e.g. IFN-*), high dose systemic steroids (e.g. ≥ 20 mg prednisone equivalent/day) for > 30 days, thalidomide, filgrastim (G-CSF), sargramostim (GM-CSF), dinitrochlorobenzene (DNCB), thymosin alpha, thymopentin, inosiplex, polyribonucleoside, ditiocarb sodium, cyclosporin, mycophenolate mofetil, methotrexate, and cancer chemotherapy.
19. No other investigational agent within 30 days of study entry
20. Any other condition which, in the opinion of the investigator, might interfere with completion of the study or evaluation of the results
21. Have active Hepatitis B virus infection (positive HBsAg) or Hepatitis C infection(defined as positive antibodies)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles E Davis, M.D., Principal Investigator — Institute of Human Virology
Locations (1):
- University of Maryland, Institute of Human Virology, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

RESULTS

PARTICIPANT FLOW:
Groups:
- 300 ug FLSC Vaccine: Highest dose vaccine group
- 150 ug FLSC Vaccine: Middle dose vaccine group
- 75 ug FLSC Vaccine: Lowest dose vaccine group
- Placebo: Placebo control group
Period: Overall Study
Arm/Group | 300 ug FLSC Vaccine | 150 ug FLSC Vaccine | 75 ug FLSC Vaccine | Placebo
Started | 18 | 16 | 15 | 16
Completed | 13 | 14 | 13 | 12
Not Completed | 5 | 2 | 2 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 3
Not completed — Lost to Follow-up | 3 | 1 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat Analysis: Subjects who received at least 1 dose of vaccine or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 ug FLSC Vaccine | 150 ug FLSC Vaccine | 75 ug FLSC Vaccine | Placebo | Total
Number analyzed (Participants) | 18 | 16 | 15 | 16 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 16 | 15 | 16 | 65
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (8.8) | 33.3 (7.2) | 36.5 (5.5) | 32.2 (7.5) | 33.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 7 | 8 | 27
  Male | 12 | 10 | 8 | 8 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2 | 4
  Not Hispanic or Latino | 17 | 16 | 14 | 14 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 8 | 11 | 11 | 43
  White | 1 | 7 | 4 | 4 | 16
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 15 | 16 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local and Systemic Reactogenicity Signs and Symptoms
Description: Signs and symptoms include pain, tenderness, maximum severity of pain and/or tenderness, erythema, induration, fever, malaise/fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and maximum severity of systemic symptoms.
Time Frame: 48 weeks
Population: Intention-to-treat Population - All subjects who received at least one dose of vaccine/placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 ug FLSC Vaccine | 150 ug FLSC Vaccine | 75 ug FLSC Vaccine | Placebo
Number analyzed (Participants) | 18 | 16 | 15 | 16
Participants
  Injection site pain | 3 | 8 | 4 | 5
  Headache | 0 | 3 | 1 | 2
  Pruritus | 1 | 1 | 1 | 2
  Nausea | 0 | 0 | 2 | 1
  Fatigue | 0 | 2 | 0 | 1
  Pyrexia | 1 | 1 | 0 | 1
  Diarrhea | 0 | 1 | 0 | 1
  Chills | 0 | 0 | 2 | 0
  Dizziness | 0 | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Related Adverse Events
Description: Treatment emergent adverse events assessed by investigator to be either possibly, probably, or definitely related to study treatment. Medical Dictionary for Regulatory Activities (MedDRA) preferred term, severity, and assessed relationship to study products.
Time Frame: 48 weeks
Population: Intention-to-treat population: Subjects who have received at least one dose of vaccine/placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 ug FLSC Vaccine | 150 ug FLSC Vaccine | 75 ug FLSC Vaccine | Placebo
Number analyzed (Participants) | 18 | 16 | 15 | 16
Participants | 7 | 9 | 7 | 8

3. Primary Outcome: Number of Participants With Sustained Decrease in CD4 Count and CD4%.
Description: CD4 count was monitored from baseline and at each study visit through study completion. Baseline CD4 and CD4% levels were calculated by taking the average of the screening and first vaccination visits. The number of individuals who had sustained (2 consecutive time points) 30% decrease in CD4 cell/ul and CD4% from baseline were counted.
Time Frame: 48 weeks
Population: The analysis included number of participants with sustained (2 consecutive time points) of 30% decrease in CD4 cell/ul and CD4%.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 ug FLSC Vaccine | 150 ug FLSC Vaccine | 75 ug FLSC Vaccine | Placebo
Number analyzed (Participants) | 18 | 16 | 15 | 16
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Binding Antibody Response Rates to FLSC
Description: Percent of participants with anti-FLSC antibodies as assessed by ELISA by 2 weeks after final vaccination
Time Frame: 2 weeks after 4th (last) vaccination.
Population: Sample size in each group was less than safety time point because of 8 volunteers who were lost to follow-up, 5 missed vaccination visits/samples, and several samples that had high background levels to individual assays.
Measure: Number; unit: percentage of participants
Arm/Group | 300 ug FLSC Vaccine | 150 ug FLSC Vaccine | 75 ug FLSC Vaccine | Placebo
Number analyzed (Participants) | 9 | 13 | 11 | 13
percentage of participants | 100 | 100 | 100 | 0

5. Secondary Outcome: Binding Antibody Response Rates to BaL-gp120
Description: Percent of participants with anti-gp120 antibodies as assessed by ELISA
Time Frame: 2 weeks after 4th (last) vaccination
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | 300 ug FLSC Vaccine | 150 ug FLSC Vaccine | 75 ug FLSC Vaccine | Placebo
Number analyzed (Participants) | 10 | 13 | 11 | 13
percentage of participants | 30 | 46 | 9 | 0

6. Secondary Outcome: Competitive Antibody Rates to CD4i Epitopes
Description: Percent of participants with antibodies competing with A32 or 17b as assessed by ELISA.
Time Frame: 2 weeks after 4th (last) vaccination
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | 300 ug FLSC Vaccine | 150 ug FLSC Vaccine | 75 ug FLSC Vaccine | Placebo
Number analyzed (Participants) | 12 | 14 | 14 | 13
percentage of participants | 100 | 100 | 64 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Placebo: Control group
Arm/Group | 300 ug FLSC Vaccine | 150 ug FLSC Vaccine | 75 ug FLSC Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 2/16 | 2/15 | 0/16
Other Adverse Events (participants affected / at risk) | 17/18 | 16/16 | 14/15 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 ug FLSC Vaccine (N=18) | 150 ug FLSC Vaccine (N=16) | 75 ug FLSC Vaccine (N=15) | Placebo (N=16)
Substance abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Substance abuse relapse resulting in hospitalization.
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Depression resulting in hospitalization
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Acute cholecystitis requiring hospitalization and surgery
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Suicidal ideation resulting in hospitalization
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Alcohol withdrawal syndrome resulting in hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 ug FLSC Vaccine (N=18) | 150 ug FLSC Vaccine (N=16) | 75 ug FLSC Vaccine (N=15) | Placebo (N=16)
Injection site pain (General disorders) | 3 (3) | 8 (13) | 4 (8) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (8) | 5 (5) | 2 (3)
Headache (Nervous system disorders) | 3 (3) | 4 (9) | 3 (4) | 1 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (7) | 2 (2) | 5 (6)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 2 (3) | 2 (4)
Fatigue (General disorders) | 2 (3) | 2 (3) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (6) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (2) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT02756208/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT02756208/ICF_001.pdf